CLINICAL TRIAL: NCT01269385
Title: Early Treatment of High Risk Chronic Lymphocytic Leukemia With Alemtuzumab, Rituximab, and PGG Beta-Glucan: A Phase I/II Trial
Brief Title: Imprime PGG, Alemtuzumab, and Rituximab in Treating Patients With High Risk Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS1084; NCI-2010-02329 (Registry Identifier: NCI-CTRP); LS1084 (Other: Mayo Clinic Cancer Center); 10-003025 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2010-12-23; First posted 2011-01-04 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2018-08

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia; Stage 0 Chronic Lymphocytic Leukemia; Stage I Chronic Lymphocytic Leukemia; Stage II Chronic Lymphocytic Leukemia
Keywords: Imprime PGG
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Alemtuzumab; Rituximab; Flow Cytometry; In Situ Hybridization, Fluorescence; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive PGG beta-glucan IV over 2-4 hours on days 1, 5, 10, 17, 24, and 31; alemtuzumab subcutaneously on days 3, 4, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33; and rituximab IV on days 10, 17, 24, and 31. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: alemtuzumab; Biological: rituximab; Drug: PGG beta-glucan; Other: flow cytometry; Other: laboratory biomarker analysis; Genetic: DNA analysis; Genetic: fluorescence in situ hybridization; Genetic: polymerase chain reaction; Genetic: polymorphism analysis; Genetic: mutation analysis

INTERVENTIONS:
Biological: alemtuzumab — Given subcutaneously
  Other Names: anti-CD52 monoclonal antibody; Campath-1H; MoAb CD52; Monoclonal Antibody Campath-1H; Monoclonal Antibody CD52
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: PGG beta-glucan — Given IV
  Other Names: Imprime PGG
Other: flow cytometry — Correlative studies
Other: laboratory biomarker analysis — Correlative studies
Genetic: DNA analysis — Correlative studies
Genetic: fluorescence in situ hybridization — Correlative studies
  Other Names: fluorescence in situ hybridization (FISH)
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR
Genetic: polymorphism analysis — Correlative studies
Genetic: mutation analysis — Correlative studies

SUMMARY:
RATIONALE: Monoclonal antibodies, such as alemtuzumab and rituximab, can kill chronic lymphocytic leukemia (CLL) cells and are effective therapies for this disease. Biological therapies, such as Imprime PGG (poly-(1-6)-beta-glucotriosyl-(1-3)-beta-glucopyranose), may stimulate the immune system in different ways and help monoclonal antibodies kill CLL cells. Giving PGG beta-glucan together with alemtuzumab and rituximab could make therapy with monoclonal antibodies, such as alemtuzumab and rituximab, more effective.

PURPOSE: This phase I/II trial is studying the side effects and best dose of PGG beta-glucan when given together with alemtuzumab and rituximab and to see how well it works in treating patients with earlier stage high-risk chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of PGG beta glucan in combination with alemtuzumab and rituximab. (Phase I) II. Assess the rate of complete response of patients with high-risk, early-intermediate stage CLL who are treated with alemtuzumab, rituximab, and PGG beta glucan before meeting standard National Cancer Institute-International Workshop on Chronic Lymphocytic Leukemia (NCI-IWCLL) criteria (Hallek, Cheson et al. 2008) for treatment. (Phase II)

SECONDARY OBJECTIVES:

I. To monitor and assess toxicity of this regimen. II. Clinical evaluation of toxicity. III. Serial monitoring of cytomegalovirus (CMV) viral load by polymerase chain reaction (PCR).

IV. To assess the rate of overall response in CLL patients using this treatment regimen.

V. To determine time to progression, time to next treatment, and duration of response in CLL patients using this treatment regimen.

TERTIARY OBJECTIVES:

I. To assess the correlation between the individual prognostic markers (17p-, 11q-, unmutated VH gene, use of VH3-21, ZAP70+, CD38+) and clinical outcome.

II. To assess response to this combination regimen using an expanded definition of response, including bone marrow studies with immunohistochemical studies for residual CLL cells and sensitive flow cytometry for minimal residual disease in patients in complete clinical remission.

OUTLINE: This is phase I, dose-escalation study of PGG beta-glucan followed by a phase II study.

Patients receive PGG beta-glucan intravenously (IV) over 2-4 hours on days 1, 5, 10, 17, 24, and 31; alemtuzumab subcutaneously (SC) on days 3, 4, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33; and rituximab IV on days 10, 17, 24, and 31. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up monthly for 3 months, every 3 months for 1 year, and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL (Hallek, Cheson et al. 2008) manifested by: Minimum threshold peripheral lymphocyte count of 5 x 10^9/L AND immunophenotypic demonstrations of a population of B lymphocytes (as defined by CD19+) which are monoclonal (light chain exclusion); CLL will be diagnosed if these cells have >= 3 of the following characteristics: CD5+, CD23+, dim surface light chain expression, dim surface CD20 expression AND fluorescence in situ hybridization (FISH) analysis is negative for IGH/CCND1 and/or immunostaining is negative for cyclin D1 expression
* >= 1 of the following poor prognosis factors: unmutated IGHV (< 2%) AND CD38 expression (>= 30% cells positive on flow cytometry); unmutated IGHV (< 2%) AND ZAP-70 expression (>= 20% cells positive on flow cytometry); use of VH3-21 gene segment irrespective of mutation status AND CD38 expression (>= 30% cells positive on flow cytometry); use of VH3-21 gene segment irrespective of mutation status AND ZAP-70 expression (>= 20% cells positive on flow cytometry); 11q22-; 17p13-
* Rai classification Stage 0, I or II that does not meet standard NCI-IWCLL criteria for treatment of CLL (Hallek, Cheson et al. 2008)
* Limited CLL disease burden with no lymph nodes > 5 cm in any diameter and splenomegaly < 6 cm below left costal margin in midclavicular line at rest
* Creatinine =< 1.5 x upper normal limit (UNL)
* Total bilirubin =< 3.0 x UNL; if total is elevated, a direct bilirubin should be performed and should be =< 1.5 x UNL
* AST =< 3.0 x UNL
* Eastern Cooperative Oncology Group (ECOG) performance status (PS): 0, 1, or 2
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Provide informed written consent
* Willing to return to a Lymphoma Specialized Program of Research Excellence (SPORE) enrolling institution for follow-up
* Willing to provide blood samples for correlative research purposes

Exclusion Criteria:

* Pregnant women
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception
* New York Heart Association Class III or IV heart disease
* Recent myocardial infarction (< 1 month)
* Uncontrolled infection
* Infection with the human immunodeficiency virus/acquired immune deficiency syndrome (HIV/AIDS), serological evidence of active hepatitis B infection (HBsAg or HBeAg positive) or positive hepatitis C serology, as further severe immunosuppression with this regimen may occur
* Evidence of active autoimmune hemolytic anemia, immune thrombocytopenia, or pure red blood cell aplasia
* Other active primary malignancy requiring treatment or limits survival to =< 2 years
* Any major surgery =< 4 weeks prior to registration
* Any previous chemotherapy or monoclonal antibody treatment for CLL
* Current use of corticosteroids; NOTE: previous corticosteroids are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-01; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Ansell, M.D., Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Dose Level 0: During one 35-day period of treatment:
  Patients receive 1 mg/kg/dose PGG (poly-(1-6)-beta-glucotriosyl-(1-3)-beta-glucopyranose) IV over 2-4 hours on days 1, 5, 10, 17, 24, and 31
  Alemtuzumab subcutaneously 3 mg day 3 10 mg day 4 30 mg days 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33;
  Rituximab 375 mg/m2 IV on days 10, 17, 24, and 31.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
- Phase I: Dose Level 1: During one 35-day period of treatment:
  Patients receive 2 mg/kg/dose PGG (poly-(1-6)-beta-glucotriosyl-(1-3)-beta-glucopyranose) IV over 2-4 hours on days 1, 5, 10, 17, 24, and 31
  Alemtuzumab subcutaneously 3 mg day 3 10 mg day 4 30 mg days 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33;
  Rituximab 375 mg/m2 IV on days 10, 17, 24, and 31.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
- Phase I: Dose Level 2; Phase II: Dose Level 2: During one 35-day period of treatment:
  Patients receive 4 mg/kg/dose PGG (poly-(1-6)-beta-glucotriosyl-(1-3)-beta-glucopyranose) IV over 2-4 hours on days 1, 5, 10, 17, 24, and 31
  Alemtuzumab subcutaneously 3 mg day 3 10 mg day 4 30 mg days 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33;
  Rituximab 375 mg/m2 IV on days 10, 17, 24, and 31.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase I: Dose Level 0 | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II: Dose Level 2
Started | 4 | 4 | 6 | 8
Completed | 3 | 3 | 6 | 8
Not Completed | 1 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients that were included in primary and secondary analyses were included in baseline information.
Groups:
- All Patients: During one 35-day period of treatment:
  Patients receive 1, 2, or 4 mg/kg/dose PGG beta-glucan IV over 2-4 hours on days 1, 5, 10, 17, 24, and 31
  Alemtuzumab subcutaneously
  3 mg day 3
  10 mg day 4
  30 mg days 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33;
  Rituximab 375 mg/m2 IV on days 10, 17, 24, and 31.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
Arm/Group | All Patients
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 61 [47 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of PGG Beta Glucan in Combination With Alemtuzumab and Rituximab Assessed by Analyzing the Number of Dose-limiting Toxicity Events (Phase I)
Description: MTD is defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients (at least 2 of a maximum of 6 new patients). A total of 6 patients treated at the MTD will be sufficient to identify common toxicities at the MTD. Three patients will be treated at a given dose level combination for at least 5 weeks to assess toxicity. If dose-limiting toxicity (DLT) is not seen in any of the 3 patients, 3 new patients will be accrued and treated at the next higher dose level. If DLT is seen in 2 or 3 of 3 patients treated at a given dose level, then the next 3 patients will be treated at the next lower dose level, if only 3 patients were enrolled and treated at this lower dose level. We tabulate the number of patients reporting a DLT.
Time Frame: First cycle of treatment (35 days)
Population: All Phase I patients that were eligible and completed cycle 1 treatment were used in the MTD assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I: Dose Level 0: During one 35-day period of treatment:
  Patients receive 1 mg/kg/dose PGG beta-glucan IV over 2-4 hours on days 1, 5, 10, 17, 24, and 31
  Alemtuzumab subcutaneously 3 mg day 3 10 mg day 4 30 mg days 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33; Rituximab 375 mg/m2 IV on days 10, 17, 24, and 31.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
- Phase I: Dose Level 1: During one 35-day period of treatment:
  Patients receive 2 mg/kg/dose PGG beta-glucan IV over 2-4 hours on days 1, 5, 10, 17, 24, and 31
  Alemtuzumab subcutaneously 3 mg day 3 10 mg day 4 30 mg days 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33;
  Rituximab 375 mg/m2 IV on days 10, 17, 24, and 31.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
- Phase I: Dose Level 2: During one 35-day period of treatment:
  Patients receive 4 mg/kg/dose PGG beta-glucan IV over 2-4 hours on days 1, 5, 10, 17, 24, and 31
  Alemtuzumab subcutaneously 3 mg day 3 10 mg day 4 30 mg days 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33;
  Rituximab 375 mg/m2 IV on days 10, 17, 24, and 31.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
Arm/Group | Phase I: Dose Level 0 | Phase I: Dose Level 1 | Phase I: Dose Level 2
Number analyzed (Participants) | 3 | 3 | 6
Participants | 0 | 0 | 1

2. Primary Outcome: Proportion of Complete Responses (Dose Level 2)
Description: The number of patients that demonstrate a Complete Response (CR) during treatment on Dose Level 2 divided by the number of eligible patients starting Dose Level 2 treatment.
  A CR requires all of the following for a period of at least 2 months: Absence of lymphadenopathy by physical examination, no hepatomegaly or splenomegaly, absence of constitutional symptoms, neutrophils >1500/ul, Platelets >100,000/ul, Hemoglobin >11.0 gm/dl, Peripheral blood lymphocytes <4000/uL.
Time Frame: 3 months after the completion of treatment, up to 5 years
Population: All patients treated at dose level 2 were included in this analysis. This includes 6 patients registered to the Phase I: Dose level 2 and 8 patients registered to Phase II.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Dose Level 2: During one 35-day period of treatment:
  Patients receive 4 mg/kg/dose PGG beta-glucan IV over 2-4 hours on days 1, 5, 10, 17, 24, and 31
  Alemtuzumab subcutaneously 3 mg day 3 10 mg day 4 30 mg days 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33;
  Rituximab 375 mg/m2 IV on days 10, 17, 24, and 31.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
Arm/Group | Dose Level 2
Number analyzed (Participants) | 14
proportion of participants | .65 [.41 to .85]

3. Secondary Outcome: Overall Response Rate (Dose Level 2)
Description: Overall response rate was estimated by the total number of patients receiving Dose Level 2 reporting complete responses or partial responses (CR or PR) divided by the total number of evaluable patients that started Dose Level 2 treatment.
  A COMPLETE RESPONSE (CR) requires all of the following for a period of at least 2 months: Absence of lymphadenopathy by physical examination, no hepatomegaly or splenomegaly, absence of constitutional symptoms, neutrophils >1500/ul, Platelets >100,000/ul, Hemoglobin >11.0 gm/dl, Peripheral blood lymphocytes <4000/uL.
  A PARTIAL RESPONSE (PR) requires the patient exhibits at least two of the features: ≥ 50% decrease in peripheral blood lymphocyte count from baseline, ≥ 50% reduction in the sum of the products of the maximal perpendicular diameters of the largest measured node or nodal masses in the right and left cervical, axillary, and inguinal lymph node regions on physical examination.
Time Frame: 3 months after the completion of treatment, up to 5 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Dose Level 2
Number analyzed (Participants) | 14
proportion of patients | .93 [.75 to 1.0]

4. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time from registration to the earliest date of documentation of disease progression. If a patient dies without a documentation of disease progression, the patient will be considered to have had tumor progression at the time of their death unless there is sufficient documented evidence to conclude no progression occurred prior to death. The distribution of time to disease progression will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 5 years
Population: All 20 eligible patients that started and completed protocol treatment were combined in this analysis to assess overall benefit of protocol treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients
Number analyzed (Participants) | 20
months | 17.6 [9.7 to 32.1]

5. Secondary Outcome: Duration of Response for All Evaluable Patients Who Have Achieved an Objective Response
Description: Duration of response is defined for all evaluable patients who have achieved an objective response as the date at which the patient's objective status is first noted to be either a CR or PR to the earliest date progression is documented. The distribution of duration of response will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 5 years
Population: Data was not collected to run this analysis.
Arm/Group | All Patients
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Subsequent Therapy
Description: Time to subsequent therapy is defined to be the time from the end of active treatment date to the date subsequent therapy is initiated. The distribution of time to subsequent therapy will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 5 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients
Number analyzed (Participants) | 20
months | NA [14.9 to NA] — Too few patients had an event (subsequent treatment) to estimate a median nor a upper 95% confidence interval.

7. Secondary Outcome: Number of Participants With Grade 3+ Adverse Events
Description: Adverse events were collected at the end of each cycle according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The number of grade 3+ events at least possibly related to treatment are recorded. For a complete set of all recorded adverse events, please see the Adverse Events section of this report.
Time Frame: up to 5 years of treatment
Population: All 20 eligible patients that started and completed protocol treatment were combined in this analysis to assess overall effect of protocol treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 20
Participants
  Grade 3 Adverse Event | 1
  Grade 4 Adverse Event | 2

ADVERSE EVENTS:
Groups:
- Dose Level 0: During one 35-day period of treatment:
  Patients receive 1 mg/kg/dose PGG beta-glucan IV over 2-4 hours on days 1, 5, 10, 17, 24, and 31
  Alemtuzumab subcutaneously 3 mg day 3, 10 mg day 4 30 mg days 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33.
  Rituximab 375 mg/m2 IV on days 10, 17, 24, and 31. Treatment continues in the absence of disease progression or unacceptable toxicity.
- Dose Level 1: During one 35-day period of treatment:
  Patients receive 2 mg/kg/dose PGG beta-glucan IV over 2-4 hours on days 1, 5, 10, 17, 24, and 31
  Alemtuzumab subcutaneously 3 mg day 3, 10 mg day 4 30 mg days 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33.
  Rituximab 375 mg/m2 IV on days 10, 17, 24, and 31. Treatment continues in the absence of disease progression or unacceptable toxicity.
- Dose Level 2: During one 35-day period of treatment:
  Patients receive 4 mg/kg/dose PGG beta-glucan IV over 2-4 hours on days 1, 5, 10, 17, 24, and 31
  Alemtuzumab subcutaneously 3 mg day 3, 10 mg day 4 30 mg days 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33.
  Rituximab 375 mg/m2 IV on days 10, 17, 24, and 31. Treatment continues in the absence of disease progression or unacceptable toxicity.
Arm/Group | Dose Level 0 | Dose Level 1 | Dose Level 2
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/4 | 4/14
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0 (N=4) | Dose Level 1 (N=4) | Dose Level 2 (N=14)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 0 (N=4) | Dose Level 1 (N=4) | Dose Level 2 (N=14)
Anemia (Blood and lymphatic system disorders) | 4 (5) | 3 (6) | 11 (40)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 4 (6)
Fever (General disorders) | 3 (5) | 2 (2) | 4 (5)
Cytokine release syndrome (Immune system disorders) | 2 (2) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 4 (5)
Lung infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (2)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (7) | 4 (13) | 14 (43)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (3) | 6 (7)
Platelet count decreased (Investigations) | 3 (5) | 3 (9) | 7 (23)
White blood cell decreased (Investigations) | 3 (3) | 2 (4) | 8 (15)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3) | 9 (11)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes